CLINICAL TRIAL: NCT00374712
Title: Study of Klotho Gene Polymorphisms in the Regulation of Serum Phosphate Levels in Hemodialysis Patients
Brief Title: Klotho Gene Polymorphism in Dialyzed Patients With Hyperphosphatemia
Status: Terminated | Type: Observational
Why Stopped: terminated
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Other Study IDs: P031010; CRC 03161
Record Dates: First submitted 2005-09-12; First posted 2006-09-11 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease; Hyperphosphatemia; Renal Osteodystrophy
Keywords: Phosphate; Dialysis; Klotho; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Hyperphosphatemia; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with chronic kidney disease (CKD) and those with end-stage renal disease (ESRD) undergoing renal replacement therapies show elevated serum phosphate levels which predispose them to cardiovascular calcifications and high risks of death from cardiovascular diseases. However, in certain patients hyperphosphatemia is not related to dialysis insufficiency, excessive daily dietary phosphorus intake or high serum parathyroid hormone (PTH) levels, suggesting that other mechanisms could be involved. Transgenic mice lacking the klotho gene showed a phenotype which resembles that of dialyzed ESRD patients, in the sense that they have hyperphosphatemia, vascular calcifications, and a short lifespan. This study will analyze whether functional polymorphisms or variants in the human klotho gene are associated with hyperphosphatemia in these patients.

DETAILED DESCRIPTION:
The entire coding region of the klotho gene will be sequenced looking for functional variants and polymorphisms that differentiate two groups of adult dialyzed ESRD patients, matched for age and gender, and with comparable values for dialysis dose and daily protein intake. These two groups consist of one group of 20 adult, dialyzed patients with serum phosphate levels > 2.50 mM compared to another group of 20 adult, dialyzed ESRD patients with serum phosphate levels < 1.50 mM. The results of this study will allow to determine whether there is a relationship between extreme hyperphosphatemia and klotho gene polymorphisms in dialysed ESRD patients.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Stable hemodialysis patients for at least 3 months
* Phosphatemia > 2.5 mM
* Kt/V > 1.2
* Total weekly phosphate removal > 75 millimoles

Group 2

* Stable hemodialysis patients for at least 3 months
* Phosphatemia < 1.5 mM
* Kt/V > 1.2
* Total weekly phosphate removal > 25 millimoles

Exclusion Criteria:

* Age > 80 years
* Insufficient dialysis dose (Kt/V < 1.2)
* Total weekly phosphate removal < 25 mM
* Problems with vascular access for hemodialysis (central catheter, arteriovenous [A-V] fistula dysfunction)
* Methods of dialysis different than the classical hemodialysis (peritoneal, hemofiltration, or hemodiafiltration with or without acetate)
* Intolerance or allergy to ARYLANE M9 dialyzers
* Hypocalcemia < 2.0 mmol/liter
* Hypophosphatemia < 0.6 mmol/liter
* Daily protein intake < 0.6 g/kg/j
* Parathyroidectomy at least 3 months prior to the study
* Evolutive neoplasia with or without secondary lytic bone lesions
* Intestinal malabsorption
* Alcoholism
* Corticotherapy
* Treatment by bisphosphonates, fluor or recombinant PTH
* Malnutrition (body mass index [BMI] < 15)
* Amputation of lower members (> 10% of total body)
* Prolonged immobilization
* Secondary hyperparathyroidism (PTH > 1400 pg/ml)
* Vitamin D deficiency (25OHD3 < 10 ng/ml)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, end-stage renal disease patients treated by standard hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2005-01; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo URENA TORRES, MD, Principal Investigator — Clinique de l'Orangerie, France
Locations (1):
- Clinique de l'Orangerie - Service de Néphrologie et Dialyse, Aubervilliers, France

REFERENCES:
- [Result] Prie D, Beck L, Urena P, Friedlander G. Recent findings in phosphate homeostasis. Curr Opin Nephrol Hypertens. 2005 Jul;14(4):318-24. doi: 10.1097/01.mnh.0000172716.41853.1e. PMID 15930998